CLINICAL TRIAL: NCT01687348
Title: Lidocaine Pharmacokinetics During Tumescent Infiltrative Anaesthesia for Mastectomy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-000817-36; 2012-05 (Other: AP HM)
Record Dates: First submitted 2012-06-20; First posted 2012-09-18 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2015-09

CONDITIONS: Mastectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lidocaine (Experimental): lidocaine traitment
  Interventions: Drug: lidocaine aguettant

INTERVENTIONS:
Drug: lidocaine aguettant

SUMMARY:
Prospective, monocentric, open-label study conducted in women requiring mastectomy and eligible for tumescent infiltrative anaesthesia.

Blood samples will be collected during 48h after start of infiltration. Total and free lidocaine concentrations measurements will be determined by gas chromatography. Visual analogic scale scores to evaluate postoperative pain and all data concerning analgesic drugs and adverse effects will be collected.

Population pharmacokinetic parameters will be estimated using NONMEM software and covariates influence on parameters variability will be tested.

Primary outcome value: Population pharmacokinetic parameters with possible covariates influence on variability.

Patients and period of study: n=30 patients enrolled during 24 months, total study duration: 30 months.

ELIGIBILITY:
Inclusion Criteria:

* Surgery carcinologique of the breast requiring a mastectomy under tumescente local anesthetic
* Age: upper to 18 years
* Weight: upper to 50 kg

Exclusion Criteria:

* Cutaneous infection in the point of draining
* Clinical Disorder(Confusion) of the coagulation
* Retreat(Withdrawal) of the consent in the course of protocol
* Unwanted Effect engraves(burns) requiring the stop(ruling) of the treatment(processing)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of 'drug lidocaine'" | 36 MONTHS
  during tumescent infiltrative anaesthesia for mastectomy.

SECONDARY OUTCOMES:
analgesic postoperative efficacy | 36 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France